CLINICAL TRIAL: NCT01502553
Title: Verify the Functions of BPM LS-802 to Comply With ANSI/AAMI SP10
Brief Title: Clinical Study of Blood Pressure Monitor in Conformance With the ANSI/AAMI SP10
Acronym: BPM_S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leo Wang (Other)
Collaborators: BTS International (Other)
Responsible Party: Sponsor-Investigator, Leo Wang, Director, BTS International
Organization: BTS International (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Trans 2011004; BTS-TRANS04 (Other: BTSInternational)
Record Dates: First submitted 2011-12-21; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Hypertension
Keywords: blood pressure; heart rate
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Pressure, Heart Rate, Monitor (Experimental): Device Comparison Test DUT: Transtek Blood Pressure Monitor, LS-802 Refrence Device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1mmHg and range: 0-300mmHg.
  Groups/Cohorts: Blood Pressure & Heart Rate Monitor
  Interventions: Device: Comparison Test to Yuyue Medical BP Meter, YYBP-212

INTERVENTIONS:
Device: Comparison Test to Yuyue Medical BP Meter, YYBP-212 — DUT: Transtek Blood Pressure Monitor, LS-802. Reference Device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1mmHg and range: 0-300mmHg.
  Other Names: Brand names: Yuyue; Serial numbers: YYBP20100013437; Code name: YYBP-212

SUMMARY:
The clinical protocol of the clinical testing of this device:

1. Objective of the test: To verify the function of device.
2. Test methods and procedures: Performance test in two positions: Seated and Supine.
3. DUT: Transtek Blood Pressure Monitor, Model: LS-802. Cuff size: 22-32 cm and 22-42 cm.
4. Comparison device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1 mmHg and range: 0-300 mmHg.
5. Study endpoints: Comply with ANSI/AAMI SP10-2002 standard.
6. Statistical methodology used: Description of statistical methods.
7. Result: Meet the requirements of SP10.

DETAILED DESCRIPTION:
Hospital Information The data was collected by Zhongshan City People's Hospital Clinical Investigator Team at Zhongshan City People's Hospital, No.2 Sunwen Dong Road, Zhongshan, Guangdong 528403, P. R. China.

Investigator: Dr. Cao Yuedong, Leader; Li Qidong, Nurse A; Chen Wenqian, Nurse B.

Contact Dr. Cao Yuedong Tel: +86 760 88823818

Used Equipments DUT (Device Under Test): Transtek Blood Pressure Monitor, Model: LS-802. Cuff size: 22-32 cm and 22-42 cm.

Reference Device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1 mmHg and range: 0-300 mmHg.

Test Protocol

1. Test Purpose:

   The aim of clinical test is to determine, for the purpose of design qualification, the overall performance of the system meeting the following requirement: For systolic and diastolic pressures, treated separately, the mean difference of the paired measurement of the test system and the comparison system shall be ± 5 mmHg or less, with standard deviation of 8 mmHg or less.
2. Target Subject:

1) The subject database shall contain at least 85 subjects. 2) The distribution of blood pressure of the subjects required to be: At least 10 percent below 100 mmHg systolic; at least 10 percent above 160 mmHg systolic; at least 10 percent below 60 mmHg diastolic; at least 10 percent above 100 mmHg diastolic; with the remainder distributed between these outer limits.

3. Identification and precision of equipment used According to ANSI/AAMI SP10, the maximum measurement error of the non-automatic sphygmomanometers used in the comparing test shall not exceed 1.0mmHg at the temperature of the test. The manometer was used to verify its accuracy before test.

The clinical study was conducted according to the protocol described in the ANSI/AAMI SP10 with 95 subjects.

4. Test procedures (auscultatory method, same-limb sequential measurement was chosen)

1. Record the age, gender, and circumference of the left arm of the subject.
2. Let subject seated or supine calmly for two minutes before test.
3. Measure heart rate in one minute by palpation on radial artery, record it.
4. As shown in Fig. 0, two observers shall make simultaneous, blinded, blood pressure determination on the subject's left arm. Each nurse will write down the reading on a small piece of paper, make a tick if there is an auscultatory gap and then submit to the recorder.
5. The two readings separately from two observers will be recorded, and if two observers agree that they find an auscultatory gap this time, it will also be recorded. The arm cuff will be take off, after 90 seconds rest, TMB-986 cuff will be taken on and tested, and the readings (systolic, diastolic, mean BP and Heart rate) be recorded.
6. For each subject, repeat 3) and 5) to get 3 measurements.
7. Repeat step 1) to 6) for every subject. 5. Note:

1) No motion and speaking are allowed during the measurement. 2) DUT uses the 22-42 cm Cuff when the arm circumference of patients above 32 cm and the other patients use 22-32 cm Cuff.

3) The reference device's cuff release at the rate about 3 mmHg/s so to ensure an accurate reading of observer.

4) The arm of the same height and heart when measurement. 5) Test environment: Temperature: 20±1 ℃; Relative humidity: 40~50%.

ELIGIBILITY:
Inclusion Criteria:

* male,female,

Exclusion Criteria:

* below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Verify the accuracy of measure functions of device | 10 days
  Verify the accuracy of device if meet the requirements of ANSI/AAMI SP10 when it measure Systolic & Diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Yuedong Cao, Doctor, Study Director — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China

REFERENCES:
- [Background] Alpert BS. Validation of the Tiba Medical Ambulo 2400 ambulatory blood pressure monitor to the ISO Standard and BHS protocol. Blood Press Monit. 2010 Oct;15(5):275-7. doi: 10.1097/MBP.0b013e32833c8b39. PMID 20559140
- See also: Related Info — http://www.zsph.com